CLINICAL TRIAL: NCT05837611
Title: Piloting Deposit Contracts to Increase Accessibility of a Contingency Management Intervention to Reduce Problematic Drinking
Brief Title: Deposit Contracts to Increase Accessibility of a Contingency Management Intervention to Reduce Problematic Drinking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of North Texas, Denton, TX (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-22
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Alcohol Abuse; Alcohol Intervention; Transdermal Alcohol Monitoring; Contingency Management; Deposit Contract
MeSH Terms: conditions — Alcoholism | interventions — Administration, Cutaneous; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monitoring Group Only (Active Comparator): Individuals in the Monitoring only group will be required to put down a 200$ deposit but will earn it back non-contingently by attending the weekly study meetings. They will be monitored using the Transdermal Alcohol Monitoring device, but will not be required to meet any Alcohol reduction goals to earn their deposit back.
  Interventions: Other: Transdermal Alcohol Monitoring
- Deposit Contract Group (Experimental): Individuals in the Deposit COntract group will be required to put down a 200$ deposit but will earn it back, as well as a bonus, contingently for meeting alcohol reduction requirements. For this study, this is counted as having a Transdermal Alcohol COntent below equal to .02 g/dl. They will be monitored using the Transdermal Alcohol Monitoring device.
  Interventions: Behavioral: Deposit Contract; Other: Transdermal Alcohol Monitoring

INTERVENTIONS:
Behavioral: Deposit Contract — A deposit contract requires individuals to put down money that is earned back contingently upon meeting their goals.
  Arms: Deposit Contract Group
Other: Transdermal Alcohol Monitoring — Using a SCRAM-Cam device participants will be monitored for their alcohol use.

SUMMARY:
This study will examine the effects of an incentive-based intervention (for reducing alcohol use) that would be sustainable, easily accessible intervention using remote alcohol monitoring and deposit contracts, targeting individuals who would not be reached by more traditional forms of treatment due to barriers such as time constraints, attitudes, and stigma.

DETAILED DESCRIPTION:
Deposit contracts are effective at treating a wide variety of problems: smoking cessation, weight loss, and increasing physical activity. Despite the promise of deposit contracts, few earlier studies targeted problem drinking, since doing so required burdensome frequent monitoring - now overcome by remote alcohol monitoring. Earlier work relied on self- and collateral reports, breath alcohol concentrations during clinic visits, or an indirect non-specific marker of alcohol use. Despite these difficulties, earlier studies of deposit contracts were encouraging, with notable increases in: therapy participation; retention ; and abstinence duration compared to previous reports. Collectively, these studies show the potential of deposit contracts to reduce problem drinking but provide only limited evidence of its effectiveness. Still, these studies, and our recent success using contingency management with remote alcohol monitoring, provide a compelling rationale for examining whether a deposit contract program might provide a feasible, effective, and accessible way of helping people reduce drinking. Though there is limited systematic research on deposit contracts, deposit contract programs for various problems are widely available and have proven quite attractive. For example, a deposit contract weight loss website, has over 887,000 users with $62M in incentives paid. However, it is unclear if deposit contracts would be acceptable (and therefore feasible) to individuals interested in reducing their problem drinking. Therefore, we feel that the proposed deposit contract intervention utilizing remote alcohol monitoring could be a widely available and acceptable intervention for problem drinking for three reasons: (1) because of the effectiveness and convenience of our contingency management intervention using remote alcohol monitoring; (2) because of the widespread success of other deposit contract programs like DietBetã; and (3) because the potentially increased attractiveness and effectiveness of an intervention that can return an amount greater than the deposit. The adoption of a deposit contract intervention plus remote alcohol monitoring will only be accelerated by the "FitBit"-style alcohol monitoring devices being developed by many companies (we are currently independently evaluating one such device). However, making deposit contracts widely available will need evidence of their effectiveness, which requires large randomized controlled trials. The purpose of this R21 application is to develop this evidence by demonstrating that deposit contracts with remote alcohol monitoring are feasible and provide evidence of effectiveness needed to design and justify future studies.

ELIGIBILITY:
Inclusion Criteria:

* at least 21 years of age
* report > 8 heavy drinking episodes during the last 28 days
* want to reduce their alcohol use
* are willing to wear a transdermal alcohol monitor
* own a smartphone
* are willing and able to deposit $200

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Transdermal Alcohol Content | 4 weeks continuously
  Measurement produced while wearing Transdermal Alcohol Monitor

CONTACTS AND LOCATIONS:
Locations (1):
- University Of North Texas, Denton, Texas, United States

REFERENCES:
- [Background] Bigelow G, Strickler D, Liebson I, Griffiths R. Maintaining disulfiram ingestion among outpatient alcoholics: a security-deposit contingency contracting procedure. Behav Res Ther. 1976;14(5):378-81. doi: 10.1016/0005-7967(76)90028-0. No abstract available. PMID 971213
- [Background] Burns RJ, Rothman AJ. Comparing Types of Financial Incentives to Promote Walking: An Experimental Test. Appl Psychol Health Well Being. 2018 Jul;10(2):193-214. doi: 10.1111/aphw.12126. Epub 2018 Apr 19. PMID 29671957
- [Background] Dallery J, Raiff BR, Grabinski MJ, Marsch LA. Technology-Based Contingency Management in the Treatment of Substance-Use Disorders. Perspect Behav Sci. 2019 Jul 9;42(3):445-464. doi: 10.1007/s40614-019-00214-1. eCollection 2019 Sep. PMID 31976444
- [Background] Ersner-Hershfield SM, Connors GJ, Maisto SA. Clinical and experimental utility of refundable deposits. Behav Res Ther. 1981;19(5):455-7. doi: 10.1016/0005-7967(81)90137-6. No abstract available. PMID 7316923
- [Background] Jarvis BP, Dallery J. Internet-based self-tailored deposit contracts to promote smoking reduction and abstinence. J Appl Behav Anal. 2017 Apr;50(2):189-205. doi: 10.1002/jaba.377. Epub 2017 Feb 17. PMID 28211949
- [Background] Paxton R. The effects of a deposit contract as a component in a behavioural programme for stopping smoking. Behav Res Ther. 1980;18(1):45-50. doi: 10.1016/0005-7967(80)90068-6. No abstract available. PMID 7369987
- [Background] Pomerleau O, Pertschuk M, Adkins D, Brady JP. A comparison of behavioral and traditional treatment for middle-income problem drinkers. J Behav Med. 1978 Jun;1(2):187-200. doi: 10.1007/BF00846639. PMID 756475
- [Background] Volpp KG, John LK, Troxel AB, Norton L, Fassbender J, Loewenstein G. Financial incentive-based approaches for weight loss: a randomized trial. JAMA. 2008 Dec 10;300(22):2631-7. doi: 10.1001/jama.2008.804. PMID 19066383
- [Background] White JS, Dow WH, Rungruanghiranya S. Commitment contracts and team incentives: a randomized controlled trial for smoking cessation in Thailand. Am J Prev Med. 2013 Nov;45(5):533-42. doi: 10.1016/j.amepre.2013.06.020. PMID 24139765